CLINICAL TRIAL: NCT04528251
Title: Comparison of the Effectiveness of Two Different Antibiotic Regimens Used in the Treatment of Pregnant Women With Preterm Rupture of Membranes Between 24 and 34 Weeks of Gestation in Preventing Neonatal Inflammation and Early Neonatal Sepsis.
Brief Title: Comparison of the Effectiveness of Two Different Antibiotic Regimens of the Treatment of Pregnant Women With Preterm Rupture of Membranes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, Principal Investigator, Hacettepe University
Other Study IDs: KA-20043
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Preterm Membrane Rupture; Neonatal Sepsis
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum IL-6, Vaginal IL-6, Vaginal PCR, Vaginal fluid direct microscopic examination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There is no consensus around the world on the treatment of preterm rupture of membranes, which is one of the important causes of early neonatal sepsis and one of the common causes of prematurity. Different countries, hospitals and physicians can determine different treatment approaches. There is very little scientific data on the benefit of commonly used treatment regimens other than experience. In this study, scientific results will be obtained by comparing the efficacy of treatments (Sulbactam ampicillin or azithromycin ampicillin) in two different hospitals (Hacettepe University Perinatology Clinic and Ankara City Hospital Perinatology Clinic), and it will be shown which treatment regimen reduces early neonatal sepsis and inflammation better. Some samples (vaginal IL-6, vaginal-cervical swab samples for atypical bacteria, cervical swab samples for direct microscopy, serum IL-6) will be taken from pregnant women who develop membrane rupture and these samples will be used as initial inflammation markers. Each physician will decide on the treatment of his own patient, there will be no intervention in the treatment of the patient within the scope of the research. Patients will continue their routine follow-up after receiving their treatment. When the delivery occurs, the level of IL-6 in the cord blood will be examined with other inflammation markers (procalcitonin, crp, complete blood count), and the neonatal inflammation status of the baby will be determined. The low inflammation markers detected in the babies of pregnant women with high initial inflammation values will be compared and it will be determined which treatment is more effective. At the same time, routine neonatal intensive care follow-ups of these babies will be continued and treatment efficiency in terms of early neonatal sepsis will be determined. This study will present scientific data on which treatment is effective in the literature and will guide international treatment guidelines. At the same time, preterm rupture of membranes will show which bacterial agent plays a more role in the etiology and which of the inflammation markers have more sensitivity and specificity, as well as the success of the treatment, which is the subject of the study. The routine use of some examinations (such as cervical PCR) performed before the treatment begins, is a guide in the selection of agent-specific treatment and may shorten the unnecessary drug use and hospital stay; The management of patients may vary according to the initial inflammation parameters. Physicians evaluating the results of this study can evaluate the risk of their babies in terms of early neonatal sepsis according to the initial inflammation values of their patients, and increase and decrease the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Having received azithromycin-ampicillin or sulbactam-ampicillin treatment during antenatal period with the diagnosis of preterm rupture of membranes that started before 34 weeks.

Exclusion Criteria:

* Having a disease detected in the perinatal or neonatal period (such as hydrops, congenital anomalies)
* Having a history of iatrogenic preterm birth
* Lethal or chromosomal anomaly
* Being diagnosed with perinatal hypoxia, hypoxic ischemic encephalopathy

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who applied to study centers with PPROM and started antibiotic treatment and their newborn babies will be included.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
maternal vaginal IL-6, vaginal-cervical swab samples for atypical bacteria, cervical swab samples for direct microscopy, serum IL-6 | 1 hour
  maternal inflammation markers
level of IL-6 in the cord blood, procalcitonin, crp, complete blood count | 1 hour
  neonatal inflammation markers

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)